CLINICAL TRIAL: NCT00549770
Title: A Multi-center, Randomized, Double-blind, Placebo and Active Controlled, Parallel Group, Dose Range Study to Evaluate the Efficacy and Safety of LCZ696 Comparatively to Valsartan, and to Evaluate AHU377 to Placebo After 8 Week Treatment in Patients With Essential Hypertension
Brief Title: Efficacy and Safety of LCZ696A in Patients With Essential Hypertension
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLCZ696A2201
Record Dates: First submitted 2007-10-05; First posted 2007-10-26 (Estimated); Results first posted 2015-08-10 (Estimated); Last update posted 2015-08-25 (Estimated); Status verified 2015-08

CONDITIONS: Hypertension
Keywords: Hypertension, valsartan, LCZ696
MeSH Terms: conditions — Hypertension | interventions — sacubitril and valsartan sodium hydrate drug combination; Valsartan; sacubitril

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (8):
- LCZ696 100 mg (Experimental): Participants received LCZ696 100 mg and matching placebo to LCZ696, Valsartan and AHU377 (5 tablets and 2 capsules) daily.
  Interventions: Drug: LCZ696; Drug: Placebo
- LCZ696 200 mg (Experimental): Participants received LCZ696 200 mg and matching placebo to LCZ696, Valsartan and AHU377 (5 tablets and 2 capsules) daily.
  Interventions: Drug: LCZ696; Drug: Placebo
- LCZ696 400 mg (Experimental): Participants received LCZ696 400 mg (200 mg LCZ696 for one week and then up-titration to 400 mg LCZ696 for 7 weeks) and matching placebo to LCZ696, Valsartan and AHU377 (5 tablets and 2 capsules) daily.
  Interventions: Drug: LCZ696; Drug: Placebo
- Valsartan 80 mg (Active Comparator): Participants received Valsartan 80 mg and matching placebo to LCZ696, Valsartan and AHU377 (5 tablets and 2 capsules) daily.
  Interventions: Drug: Valsartan; Drug: Placebo
- Valsartan 160 mg (Active Comparator): Participants received Valsartan 160 mg and matching placebo to LCZ696, Valsatan and AHU377 (5 tablets and 2 capsules) daily.
  Interventions: Drug: Valsartan; Drug: Placebo
- Valsartan 320 mg (Active Comparator): Participants received Valsartan 320 mg (160 mg valsartan capsules for one week followed by 320 mg valsartan capsules for 7 weeks) and matching placebo to LCZ696, Valsartan and AHU377 (5 tablets and 2 capsules) daily.
  Interventions: Drug: Valsartan; Drug: Placebo
- AHU377 200 mg (Experimental): Participants received AHU377 200 mg and matching placebo to LCZ696 and Valsartan (5 tablets and 2 capsules) daily.
  Interventions: Drug: AHU377; Drug: Placebo
- Placebo (Placebo Comparator): Participants received matching placebo to LCZ696, Valsartan and AHU377 (5 tablets and 2 capsules) daily.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LCZ696
  Arms: LCZ696 100 mg; LCZ696 200 mg; LCZ696 400 mg
Drug: Valsartan
  Arms: Valsartan 160 mg; Valsartan 320 mg; Valsartan 80 mg
Drug: AHU377
  Arms: AHU377 200 mg
Drug: Placebo

SUMMARY:
This study was a dose-ranging efficiacy study in patients with essential hypertension to assess the blood pressure lowering effect, and safety of LCZ696 compared to valsartan and placebo. The study will also evaluate the efficacy and safety of AHU377 as compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Male or females from 18 up to and including 75 years
* Patients with mild-to-moderate uncomplicated essential hypertension, untreated or currently taking antihypertensive therapy (monotherapy or combination therapy of 2 drugs; therapy with a fixed dose combination of two active substances represents 2 drugs)
* Untreated patients must have had an office msDBP≥ 95 mmHg at the randomization visit (Visit 3) and the 2 preceding visits (Visits 1 and 2).
* Treated patients must have had an office msDBP≥ 90 mmHG after washout (Visit 2), and a msDBP> 95 mmHg at baseline (Visit 3);

Exclusion Criteria:

* Severe hypertension (msSBP ≥180 mmHg and/or msDBP ≥110 mmHg)
* History of angioedema, drug-related or otherwise, as reported by the patient
* Type 1 or Type 2 diabetes mellitus (according to the ADA criteria)
* History or evidence of a secondary form of hypertension, such as renal parenchymal hypertension, renovascular hypertension, coarctation of the aorta, primary hyperaldosteronism, Cushing's disease, drug-induced hypertension, unilateral or bilateral renal artery stenosis, pheochromocytoma, polycystic kidney disease, etc.
* History of angina pectoris, myocardial infarction, coronary bypass surgery, ischemic heart disease, surgical or percutaneous arterial intervention of any kind (coronary, carotid or peripheral intervention), stroke, TIA (transient ischemic attack), carotid artery stenosis, aortic aneurysm or peripheral arterial disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1334 (Actual)
Dates: Start 2007-09; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals; Novartis Pharmaceuticals, Study Chair — Novartis Pharmaceuticals
Locations (159):
- United States (33):
  - Novartis Investigative Site, Birmingham, Alabama
  - Novartis Investigative Site, Muscle Shoals, Alabama
  - Novartis Investigative Site, Chandler, Arizona
  - Novartis Investigative Site, Buena Park, California
  - Novartis Investigative Site, Fair Oaks, California
  - Novartis Investigative Site, Long Beach, California
  - Novartis Investigative Site, Los Angeles, California
  - Novartis Investigative Site, Orangevale, California
  - Novartis Investigative Site, Santa Ana, California
  - Novartis Investigative Site, Stockton, California
  - Novartis Investigative Site, Tustin, California
  - Novartis Investigative Site, Jacksonville, Florida
  - Novartis Investigative Site, Pembroke Pines, Florida
  - Novartis Investigative Site, Pensacola, Florida
  - Novartis Investigative Site, Augusta, Georgia
  - Novartis Investigative Site, Chicago, Illinois
  - Novartis Investigative Site, Peoria, Illinois
  - Novartis Investigative Site, Baton Rouge, Louisiana
  - Novartis Investigative Site, Metairie, Louisiana
  - Novartis Investigative Site, Chelsea, Michigan
  - Novartis Investigative Site, Royal Oak, Michigan
  - Novartis Investigative Site, Brooklyn Center, Minnesota
  - Novartis Investigative Site, City of Saint Peters, Missouri
  - Novartis Investigative Site, Toms River, New Jersey
  - Novartis Investigative Site, Trenton, New Jersey
  - Novartis Investigative Site, Cincinnati, Ohio
  - Novartis Investigative Site, Oklahoma City, Oklahoma
  - Novartis Investigative Site, Simpsonville, South Carolina
  - Novartis Investigative Site, Dallas, Texas
  - Novartis Investigative Site, Houston, Texas
  - Novartis Investigative Site, Lake Jackson, Texas
  - Novartis Investigative Site, Richmond, Virginia
  - Novartis Investigative Site, Charleston, West Virginia
- Argentina (3):
  - Novartis Investigative Site, Caba, Buenos Aires
  - Novartis Investigative Site, Corrientes, Corrientes Province
  - Novartis Investigative Site, Rosario, Santa Fe Province
- Canada (9):
  - Novartis Investigative Site, Cambridge, Ontario
  - Novartis Investigative Site, Mississauga, Ontario
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Granby, Quebec
  - Novartis Investigative Site, Longueil, Quebec
  - Novartis Investigative Site, Montreal, Quebec
  - Novartis Investigative Site, Sherbrooke, Quebec
  - Novartis Investigative Site, Ste-Foy, Quebec
  - Novartis Investigative Site, Saskatoon, Saskatchewan
- Denmark (7):
  - Novartis Investigative Site, Aalborg
  - Novartis Investigative Site, Aalborg SV
  - Novartis Investigative Site, Espergærde
  - Novartis Investigative Site, Greve
  - Novartis Investigative Site, Roslev
  - Novartis Investigative Site, Vaerloese
  - Novartis Investigative Site, Viborg
- Finland (4):
  - Novartis Investigative Site, Helsinki
  - Novartis Investigative Site, Kerava
  - Novartis Investigative Site, Oulu
  - Novartis Investigative Site, Tampere
- France (8):
  - Novartis Investigative Site, Bourges
  - Novartis Investigative Site, La Chapelle-sur-Erdre
  - Novartis Investigative Site, La Roche-sur-Yon
  - Novartis Investigative Site, Le Pradet
  - Novartis Investigative Site, Murs Erigné
  - Novartis Investigative Site, Saint-Avertin
  - Novartis Investigative Site, Tours
  - Novartis Investigative Site, Vihiers
- Germany (17):
  - Novartis Investigative Site, Balve
  - Novartis Investigative Site, Beckingen
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Einbeck
  - Novartis Investigative Site, Erfurt
  - Novartis Investigative Site, Giengen an der Brenz
  - Novartis Investigative Site, Hagen
  - Novartis Investigative Site, Haigerloch
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Kassel
  - Novartis Investigative Site, Krefeld
  - Novartis Investigative Site, Mahlberg
  - Novartis Investigative Site, Messkirch
  - Novartis Investigative Site, Reinfeld
  - Novartis Investigative Site, Siegen
  - Novartis Investigative Site, Wallerfing
  - Novartis Investigative Site, Warendorf
- Hungary (4):
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Esztergom
  - Novartis Investigative Site, Miskolc
  - Novartis Investigative Site, Nyiregyháza
- Italy (16):
  - Novartis Investigative Site, Caserta, CE
  - Novartis Investigative Site, Cona, FE
  - Novartis Investigative Site, Florence, FI
  - Novartis Investigative Site, Pozzilli, IS
  - Novartis Investigative Site, Rozzano, MI
  - Novartis Investigative Site, Vimercate, MI
  - Novartis Investigative Site, Palermo, PA
  - Novartis Investigative Site, Padua, PD
  - Novartis Investigative Site, Pisa, PI
  - Novartis Investigative Site, Casorate Primo, PV
  - Novartis Investigative Site, Pavia, PV
  - Novartis Investigative Site, Stradella, PV
  - Novartis Investigative Site, Mercato San Severino, SA
  - Novartis Investigative Site, Sassari, SS
  - Novartis Investigative Site, San Daniele del Friuli, UD
  - Novartis Investigative Site, Vibo Valentia, VV
- Latvia (4):
  - Novartis Investigative Site, Daugavplis
  - Novartis Investigative Site, Kuldīga
  - Novartis Investigative Site, Ogre
  - Novartis Investigative Site, Riga
- Lithuania (3):
  - Novartis Investigative Site, Alytus
  - Novartis Investigative Site, Kaunas
  - Novartis Investigative Site, Klaipėda
- Netherlands (9):
  - Novartis Investigative Site, 's-Hertogenbosch
  - Novartis Investigative Site, Deurne
  - Novartis Investigative Site, Ermelo
  - Novartis Investigative Site, Hoogwoud
  - Novartis Investigative Site, Leeuwarden
  - Novartis Investigative Site, Losser
  - Novartis Investigative Site, Oude Pekela
  - Novartis Investigative Site, Poortvliet
  - Novartis Investigative Site, Wamel
- Poland (3):
  - Novartis Investigative Site, Ostrów Wielkopolski
  - Novartis Investigative Site, Oława
  - Novartis Investigative Site, Tarnów
- Russia (3):
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, S.-Petersburg
  - Novartis Investigative Site, Saint Petersburg
- Slovakia (6):
  - Novartis Investigative Site, Banská Bystrica, Slovak Republic
  - Novartis Investigative Site, Bratislava, Slovak Republic
  - Novartis Investigative Site, Nitra, Slovak Republic
  - Novartis Investigative Site, Prešov, Slovak Republic
  - Novartis Investigative Site, Dunajská Streda
  - Novartis Investigative Site, Žilina
- Spain (17):
  - Novartis Investigative Site, Seville, Andalusia
  - Novartis Investigative Site, Palma de Mallorca, Balearic Islands
  - Novartis Investigative Site, Badalona, Catalonia
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Tàrrega, Catalonia
  - Novartis Investigative Site, Vic, Catalonia
  - Novartis Investigative Site, Begonte, Galicia
  - Novartis Investigative Site, Santiago de Compostela, Galicia
  - Novartis Investigative Site, Madrid, Madrid
  - Novartis Investigative Site, Alicante, Valencia
  - Novartis Investigative Site, Benidorm, Valencia
  - Novartis Investigative Site, Quart de Poblet, Valencia
  - Novartis Investigative Site, Valencia, Valencia
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Hospitalet de Llbregat
  - Novartis Investigative Site, Petrel
  - Novartis Investigative Site, Riudecols
- Sweden (7):
  - Novartis Investigative Site, Boden, Sweden
  - Novartis Investigative Site, Skellefteå, Sweden
  - Novartis Investigative Site, Arvidsjaur
  - Novartis Investigative Site, Karlstad
  - Novartis Investigative Site, Kil
  - Novartis Investigative Site, Kristianstad
  - Novartis Investigative Site, Lund
- Taiwan (6):
  - Novartis Investigative Site, Taipei, Taiwan
  - Novartis Investigative Site, Taichung, Taiwan ROC
  - Novartis Investigative Site, Tainan, Taiwan ROC
  - Novartis Investigative Site, Changhua
  - Novartis Investigative Site, Taichung County
  - Novartis Investigative Site, Taipei

REFERENCES:
- [Derived] Andersen MB, Simonsen U, Wehland M, Pietsch J, Grimm D. LCZ696 (Valsartan/Sacubitril)--A Possible New Treatment for Hypertension and Heart Failure. Basic Clin Pharmacol Toxicol. 2016 Jan;118(1):14-22. doi: 10.1111/bcpt.12453. Epub 2015 Sep 4. PMID 26280447
- [Derived] Ruilope LM, Dukat A, Bohm M, Lacourciere Y, Gong J, Lefkowitz MP. Blood-pressure reduction with LCZ696, a novel dual-acting inhibitor of the angiotensin II receptor and neprilysin: a randomised, double-blind, placebo-controlled, active comparator study. Lancet. 2010 Apr 10;375(9722):1255-66. doi: 10.1016/S0140-6736(09)61966-8. Epub 2010 Mar 16. PMID 20236700

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study comprised 3 periods: a 4-week washout and placebo run-in period (pre-randomization), an 8-week randomized, double-blind monotherapy period, and 1-week randomized, placebo-controlled withdrawal period. In the randomized withdrawal, participants were either randomized to placebo or continued their original assigned treatment.
Pre-assignment Details: After successful completion of the pre-randomization period, participants were randomized 1:1:1:1:1:1:1:1 ratio to one of 8 treatment groups.
Groups:
- Valsartan 160 mg: Participants received Valsartan 160 mg and matching placebo to LCZ696, Valsartan and AHU377 (5 tablets and 2 capsules) daily.
Period: Overall Study
Arm/Group | LCZ696 100 mg | LCZ696 200 mg | LCZ696 400 mg | Valsartan 80 mg | Valsartan 160 mg | Valsartan 320 mg | AHU377 200 mg | Placebo
Started | 156 | 169 | 172 | 163 | 166 | 164 | 165 | 173
Intent-to-treat Population | 154 | 168 | 170 | 163 | 163 | 163 | 164 | 172
Ambulatory Blood Pressure Monitoring | 48 | 61 | 53 | 55 | 49 | 54 | 50 | 57
Completed | 149 | 158 | 162 | 147 | 149 | 151 | 151 | 148
Not Completed | 7 | 11 | 10 | 16 | 17 | 13 | 14 | 25
Not completed — Protocol deviation | 1 | 1 | 1 | 2 | 2 | 2 | 1 | 2
Not completed — Administrative problems | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 2 | 2 | 3 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 4 | 6 | 4 | 5 | 6 | 6 | 4 | 9
Not completed — Lack of Efficacy | 1 | 0 | 2 | 3 | 5 | 1 | 3 | 8
Not completed — Abnormal test procedure results | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 1
Not completed — Abnormal laboratory values | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Adverse Event | 1 | 3 | 1 | 2 | 1 | 0 | 5 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LCZ696 100 mg | LCZ696 200 mg | LCZ696 400 mg | Valsartan 80 mg | Valsartan 160 mg | Valsartan 320 mg | AHU377 200 mg | Placebo | Total
Number analyzed (Participants) | 156 | 169 | 172 | 163 | 166 | 164 | 165 | 173 | 1328
Age, Continuous [Mean (Standard Deviation); unit: years] | 53 (10.4) | 54 (9.7) | 52 (10.9) | 53 (9.6) | 53 (9.7) | 53 (10.1) | 53 (10.7) | 54 (10.6) | 53 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61 | 77 | 75 | 68 | 68 | 65 | 75 | 79 | 568
  Male | 95 | 92 | 97 | 95 | 98 | 99 | 90 | 94 | 760

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Mean Sitting Diastolic Blood Pressure (msDBP)
Description: Sitting BP measurements were performed at screening through the end of the study at every study visit. A negative change from baseline indicates improvement.
Time Frame: baseline, week 8
Population: Intent-to-treat (ITT): The ITT included all randomized participants who had a baseline and at least one post-baseline efficacy measuremet during the 8-week core treatment period.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | LCZ696 100 mg | LCZ696 200 mg | LCZ696 400 mg | Valsartan 80 mg | Valsartan 160 mg | Valsartan 320 mg | AHU377 200 mg | Placebo
Number analyzed (Participants) | 154 | 168 | 170 | 163 | 163 | 163 | 164 | 172
mmHg | -9.97 (0.73) | -12.92 (0.70) | -13.63 (0.70) | -9.14 (0.72) | -9.95 (0.71) | -10.93 (0.71) | -9.76 (0.71) | -6.78 (0.69)

2. Secondary Outcome: Change From Baseline in Mean Sitting Systolic Blood Pressure (msSBP)
Description: Sitting BP measurements were performed at screening through the end of the study at every study visit.
Time Frame: baseline, week 8
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | LCZ696 100 mg | LCZ696 200 mg | LCZ696 400 mg | Valsartan 80 mg | Valsartan 160 mg | Valsartan 320 mg | AHU377 200 mg | Placebo
Number analyzed (Participants) | 154 | 168 | 170 | 163 | 163 | 163 | 164 | 172
mmHg | -13.75 (1.15) | -18.70 (1.10) | -20.17 (1.10) | -12.44 (1.12) | -13.42 (1.12) | -14.16 (1.12) | -11.93 (1.11) | -7.72 (1.09)

3. Secondary Outcome: Change From Baseline in 24-hour Mean Ambulatory DBP (maDBP) and maSBP
Description: Hourly mean ambulatory DBP and SBP post-dosing was calculated for each post-dosing hour over 24 hours by taking the average of the readings taken in the corresponding post-dosing hour at randomization and at week 8.
Time Frame: baseline, 8 weeks
Population: Ambulatory Blood Pressure Monitoring (ABPM) Subset: The ABPM subest included all ITT participants who had both baseline and week 8 ABPM values.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | LCZ696 100 mg | LCZ696 200 mg | LCZ696 400 mg | Valsartan 80 mg | Valsartan 160 mg | Valsartan 320 mg | AHU377 200 mg | Placebo
Number analyzed (Participants) | 48 | 61 | 53 | 55 | 49 | 54 | 50 | 57
mmHg
  maDBP | -3.80 (0.72) | -6.78 (0.64) | -8.32 (0.71) | -4.56 (0.67) | -6.25 (0.70) | -7.13 (0.67) | -3.67 (0.70) | -1.33 (0.67)
  maSBP | -7.80 (1.04) | -11.50 (0.93) | -14.56 (1.03) | -7.29 (0.96) | -8.27 (1.00) | -9.42 (0.97) | -5.18 (1.02) | -2.90 (0.96)

4. Secondary Outcome: Change From Baseline in Daytime maDBP and maSBP
Description: Hourly mean ambulatory DBP and SBP post-dosing was calculated for each post-dosing hour over 24 hours by taking the avergae of the readings taken in the corresponding post-dosing hour at randomization and at week 8. Daytime mean SBP and DBP were the averages of the hourly means between 6 am and 10 pm.
Time Frame: baseline, 8 weeks
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | LCZ696 100 mg | LCZ696 200 mg | LCZ696 400 mg | Valsartan 80 mg | Valsartan 160 mg | Valsartan 320 mg | AHU377 200 mg | Placebo
Number analyzed (Participants) | 48 | 61 | 53 | 55 | 49 | 54 | 50 | 57
mmHg
  maDBP | -4.05 (1.23) | -6.91 (1.12) | -7.80 (1.19) | -4.78 (1.17) | -7.40 (1.23) | -7.47 (1.17) | -3.18 (1.22) | -1.53 (1.14)
  maSBP | -7.96 (1.73) | -11.76 (1.58) | -14.20 (1.67) | -7.59 (1.65) | -9.54 (1.73) | -9.90 (1.66) | -4.49 (1.72) | -3.40 (1.61)

5. Secondary Outcome: Change From Baseline in Nighttime maDBP and maSBP
Description: Hourly mean ambulatory DBP and SBP post-dosing was calculated for each post-dosing hour over 24 hours by taking the average of the readings taken in the corresponding post-dosing hour at randomization and at week 8. Nighttime mean SBP and DBP were the averages of the hourly means between 10 pm and 6 am.
Time Frame: baseline, 8 weeks
Population: Participants from the ABPM subset, who had both baseline nighttime and week 8 nighttime values, were included in the analysis only.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | LCZ696 100 mg | LCZ696 200 mg | LCZ696 400 mg | Valsartan 80 mg | Valsartan 160 mg | Valsartan 320 mg | AHU377 200 mg | Placebo
Number analyzed (Participants) | 45 | 59 | 47 | 54 | 48 | 53 | 47 | 55
mmHg
  maDBP | -2.87 (1.25) | -7.73 (1.13) | -6.93 (1.23) | -4.04 (1.17) | -4.18 (1.24) | -6.17 (1.18) | -3.31 (1.24) | -1.01 (1.16)
  maSBP | -6.40 (1.77) | -11.85 (1.60) | -12.04 (1.73) | -6.43 (1.66) | -5.82 (1.74) | -7.51 (1.67) | -3.99 (1.75) | -2.09 (1.63)

6. Secondary Outcome: Percentage of Participants Who Achieved a Successful Response in msDBP
Description: Successful response in msDBP is defined as msDBP <90 mmHg or a reduction ≥ 10 mmHg from baseline.
Time Frame: 8 weeks
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | LCZ696 100 mg | LCZ696 200 mg | LCZ696 400 mg | Valsartan 80 mg | Valsartan 160 mg | Valsartan 320 mg | AHU377 200 mg | Placebo
Number analyzed (Participants) | 154 | 168 | 170 | 163 | 163 | 163 | 164 | 172
Percentage of participants | 53.90 | 69.64 | 74.12 | 51.53 | 55.83 | 63.19 | 54.27 | 39.53

7. Secondary Outcome: Percentage of Participants Who Achieved a Successful Response in msSBP
Description: Successful response in msSBP is defined as msSBP <140 mmHg or a reduction ≥ 20 mmHg from baseline.
Time Frame: 8 weeks
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | LCZ696 100 mg | LCZ696 200 mg | LCZ696 400 mg | Valsartan 80 mg | Valsartan 160 mg | Valsartan 320 mg | AHU377 200 mg | Placebo
Number analyzed (Participants) | 154 | 168 | 170 | 163 | 163 | 163 | 164 | 172
Percentage of participants | 55.84 | 63.69 | 72.35 | 51.53 | 51.53 | 57.06 | 46.34 | 37.79

8. Secondary Outcome: Percentage of Participants Who Achieved Successful Control in msDBP
Description: Successful control in msDBP is defined as msDBP <90 mmHg.
Time Frame: 8 weeks
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | LCZ696 100 mg | LCZ696 200 mg | LCZ696 400 mg | Valsartan 80 mg | Valsartan 160 mg | Valsartan 320 mg | AHU377 200 mg | Placebo
Number analyzed (Participants) | 154 | 168 | 170 | 163 | 163 | 163 | 164 | 172
Percentage of participants | 47.40 | 60.12 | 65.88 | 45.40 | 47.85 | 56.44 | 46.95 | 38.37

9. Secondary Outcome: Percentage of Participants Who Achieved Successful Control in msSBP
Description: Successful control in msSBP is defined as <140 mmHg.
Time Frame: 8 weeks
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | LCZ696 100 mg | LCZ696 200 mg | LCZ696 400 mg | Valsartan 80 mg | Valsartan 160 mg | Valsartan 320 mg | AHU377 200 mg | Placebo
Number analyzed (Participants) | 154 | 168 | 170 | 163 | 163 | 163 | 164 | 172
Percentage of participants | 47.40 | 56.55 | 62.94 | 45.40 | 42.33 | 53.37 | 37.20 | 31.98

ADVERSE EVENTS:
Arm/Group | LCZ696 100 mg | LCZ696 200 mg | LCZ696 400 mg | Valsartan 80 mg | Valsartan 160 mg | Valsartan 320 mg | AHU377 200 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 1/156 | 0/169 | 1/172 | 1/163 | 0/166 | 0/164 | 0/165 | 0/173
Other Adverse Events (participants affected / at risk) | 4/156 | 4/169 | 4/172 | 5/163 | 4/166 | 3/164 | 5/165 | 13/173
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LCZ696 100 mg (N=156) | LCZ696 200 mg (N=169) | LCZ696 400 mg (N=172) | Valsartan 80 mg (N=163) | Valsartan 160 mg (N=166) | Valsartan 320 mg (N=164) | AHU377 200 mg (N=165) | Placebo (N=173)
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LCZ696 100 mg (N=156) | LCZ696 200 mg (N=169) | LCZ696 400 mg (N=172) | Valsartan 80 mg (N=163) | Valsartan 160 mg (N=166) | Valsartan 320 mg (N=164) | AHU377 200 mg (N=165) | Placebo (N=173)
Headache (Nervous system disorders) | 4 | 4 | 4 | 5 | 4 | 3 | 5 | 13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other